CLINICAL TRIAL: NCT06402058
Title: A Randomized, Subject and Evaluator Blinded, Matched Pairs, Pilot Study to Evaluate the Safety and Efficacy of DMSB01 According to the Number of Injections in Subjects With Crow's Feet Lines Compared to Control Device
Brief Title: A Study Comparing DMSB01 and Rejuran® for Temporary Crow's Feet Lines Improvement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMSB01_CF_301
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Crow's Feet Lines

STUDY DESIGN:
Intervention Model Description: A Randomized, Subject and Evaluator blinded, Matched pairs, Pilot Study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DMSB01 (Experimental): mPEG-PLA
  Interventions: Device: DMSB01
- Rejuran® (Active Comparator): PN
  Interventions: Device: Rejuran®

INTERVENTIONS:
Device: DMSB01 — Apply a maximum of 1.0 ml for each side of the Crow's Feet Lines using both the test device (DMSB01) and the control device (Rejuran®).
  Arms: DMSB01
Device: Rejuran® — Apply a maximum of 1.0 ml for each side of the Crow's Feet Lines using both the test device (DMSB01) and the control device (Rejuran®).
  Arms: Rejuran®

SUMMARY:
The objective of this Pilot Study is to verify the safety and efficacy of DMSB01 in the temporary improvement of Crow's Feet Lines

ELIGIBILITY:
Inclusion Criteria:

1. Among those who desire improvement in both sides of the crow's feet and have a Crow's Feet Grading Scale (CFGS) score of 2 or higher for both relaxed and maximum smile conditions
2. Individuals who have consented to abstain from any other dermatological procedures or treatments, including treatments for wrinkle reduction in the facial area, during the duration of this study

Exclusion Criteria:

1. Individuals with abnormal findings in visual-related tests (visual acuity test, Confrontational visual fields test, ocular motility test), specifically those with low vision (best-corrected visual acuity of 0.3 or less in the better eye).
2. Individuals who need to take anticoagulants from 2 weeks before the application of the investigational medical device to 2 weeks after the final application (with the exception of low dosage aspirin 100mg (up to a maximum of 300mg/day))
3. Individuals who need to take Vitamin E preparations, NSAIDs, or collagen preparations from 1 week before the application of the investigational medical device to 1 week after the final application.
4. History of bleeding disorder in past or present

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-10 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in CFGS at 4, 8, 12 weeks after the last application of the clinical trial medical device compared to the baseline evaluated by Investigator and independent evaluators | 4, 8, 12 weeks
  The Crow's Feet Grading Scale is a 5-point scale with 0 = Absent; 1 = Mild; 2 = Moderate; 3 = Severe and 4 = Extreme. 0 is the best outcome while 4 is the worst outcome. The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jongho Kim, M.D.,Ph.D., Principal Investigator — Seoul National University Bundang Hospital